CLINICAL TRIAL: NCT05888571
Title: A Randomized Controlled Trial of Prepectoral Breast Reconstruction With and Without Mesh
Brief Title: Pre-pectoral Breast Reconstruction With or Without Mesh
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20230013
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-05

CONDITIONS: Prepectoral Breast Reconstruction; TiLOOP Mesh

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prepectoral breast reconstruction with Mesh (Active Comparator): Immediate prepectoral breast reconstruction with Mesh
  Interventions: Procedure: prepectoral breast reconstruction; Procedure: Tiloop Mesh implantation
- prepectoral breast reconstruction without Mesh (Experimental): Immediate prepectoral breast reconstruction without Mesh
  Interventions: Procedure: prepectoral breast reconstruction

INTERVENTIONS:
Procedure: prepectoral breast reconstruction — Patients receive immediate prepectoral breast reconstruction
Procedure: Tiloop Mesh implantation — Patients receive immediate prepectoral breast reconstruction with Tiloop Mesh
  Arms: prepectoral breast reconstruction with Mesh

SUMMARY:
To explore the efficacy and safety that occur after immediate prepectoral breast reconstruction when TiLOOP Mesh is used compared to that when TiLOOP Mesh is not used.

DETAILED DESCRIPTION:
The clinical study aims to explore the efficacy and safety that occur after immediate prepectoral breast reconstruction when TiLOOP Mesh is used compared to that not using TiLOOP Mesh.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women aged 18-65 years who plan to undergo unilateral or bilateral immediate prepectoral prothesis breast reconstruction;
2. SSM or NSM or Skin-Reducing Mastectomy for breast cancer patients or prophylactic mastectomy;
3. Tissue expander size =<800cc, implant size =<600cc;
4. The blood perfusion of breast skin flap was well;
5. Do not smoking in the last 4 weeks or more
6. Patients with normal expectations and mental health for breast reconstruction;
7. Signed consent to participate

Exclusion Criteria:

1. Poor perfusion of breast mastectomy flap;
2. II stage breast reconstruction patients;
3. History of chest radiotherapy;
4. BMI greater than 35;
5. Patients who have not quit smoking within the last 4 weeks;

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Major Complication Rates | up to 12 months after surgery
  The rate of major complications in the two groups
Patient Breast-Q questionnaire | up to 12 months after surgery
  We use the Breast-Q questionnaire to evaluate patients' satisfaction via the reconstruction module of BREAST-Q.

SECONDARY OUTCOMES:
Minor Complication Rates | up to 12 months after surgery
  The rate of minor complications in the two groups
Rates of capsule contracture | up to 24 months after surgery
  The rates of capsule contracture in the two groups
The rate of surgical revision of reconstructed breasts | up to 12 months after surgery
  To record the rate of surgical revision events of the reconstructed breasts
The rate of implant or tissue expander removal | up to 12 months after surgery
  The rate of implant or tissue expander removal in the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No